CLINICAL TRIAL: NCT05878561
Title: A Randomized, Double-blind, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of BR1015 Combination Therapy in Comparison With Fimasartan Monotherapy for Essential Hypertension Patients Not Adequately Responded by Fimasartan 30 mg
Brief Title: A Study to Evaluate the Efficacy and Safety of BR1015 Combination Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FIC-CT-301
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan; Indapamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fimasartan + Indapamide (Experimental): Treatment Period I, II
  Interventions: Drug: Fimasartan + Indapamide
- Fimasartan + Indapamide placebo (Active Comparator): Treatment Period I, II
  Interventions: Drug: Fimasartan + Indapamide placebo

INTERVENTIONS:
Drug: Fimasartan + Indapamide — a fixed dose combination
  Other Names: I : BR1015-3 + BR1015-2, II : BR1015-1 + BR1015-2
  Arms: Fimasartan + Indapamide
Drug: Fimasartan + Indapamide placebo — a fixed dose combination
  Other Names: I : BR1015-3 + BR1015-4, II : BR1015-1 + BR1015-4
  Arms: Fimasartan + Indapamide placebo

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of BR1015 Combination therapy group in comparison with Fimasartan monotherapy group at Week 8 for essential hypertension patients who do not adequately responded by Fimasartan 30 mg

ELIGIBILITY:
* Inclusion Criteria:

  * Patients with uncontrolled essential hypertension at screening(V1) under the following criteria:

    * Naïve : 140 mmHg ≤ SiSBP < 180 mmHg
    * Use antihypertensive drugs : 130 mmHg ≤ SiSBP < 180 mmHg
  * Patients with uncontrolled essential hypertension at randomization(V2) after Fimasartan 30mg monotherapy for 4 weeks under the following criteria:

    * Selected reference arm : 140 mmHg ≤ SiSBP < 180 mmHg (For patients with cardiovascular disease, diabetes or chronic kidney disease (CKD) with albuminuria, 130 mmHg ≤ SiSBP < 180 mmHg)
    * Treatment compliance of Fimasartan 30 mg ≥70% at baseline visit (V2)
  * Voluntarily provided a written consent to participate in this clinical study
  * Able to understand this study, be cooperative in the execution of the study, and participate in the study until its completion
* Exclusion Criteria:

  * Patients taking three or more antihypertensive drugs of different families
  * Patients with blood pressure results showing SiSBP ≥ 180 mmHg or SiDBP ≥ 110 mmHg in the selected reference arm at screening(V1) and randomization(V2)
  * Patients with a difference of SiSBP ≥ 20 mmHg and SiDBP ≥ 10 mmHg in blood pressure measured three times on both arms at screening(V1)
  * Patients with secondary hypertension: Secondary hypertension is not limited to the following diseases; (e.g., coarctation of the aorta, Primary hyperaldosteronism, renal artery stenosis, Cushing's syndrome, pheochromocytoma and polycystic kidney disease, etc.)
  * Patients with orthostatic hypotension accompanied by symptoms
  * Patients who need to be administered in combination with antihypertensive drugs other than investigational product while participating in clinical trials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Sitting systolic blood pressure | 8weeks from Baseline Visit
  The change of sitting systolic blood pressure

SECONDARY OUTCOMES:
Sitting systolic blood pressure | 4weeks from Baseline Visit
  The change of sitting systolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Bucheon St.Mary's Hospital, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No